CLINICAL TRIAL: NCT05364177
Title: Comparison of 68Ga-pentixather and 68Ga-pentixafor PET/CT in Patients With Multiple Myeloma
Brief Title: 68Ga-pentixather and 68Ga-pentixafor PET/CT in Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-MM-pentixather
Record Dates: First submitted 2021-11-10; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; CXCR4; 68Ga-pentixather; PET/CT; 68Ga-pentixafor
MeSH Terms: conditions — Multiple Myeloma | interventions — 68Ga-pentixafor

STUDY DESIGN:
Intervention Model Description: 68Ga-pentixather PET/CT, 68Ga-pentixafor PET/CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-pentixather PET/CT and 68Ga-pentixafor PET/CT scan (Experimental): Participants with multiple myeloma will perform 68Ga-pentixather PET/CT and 68Ga-pentixafor PET/CT within 7-day interval
  Interventions: Drug: 68Ga-Pentixather; Drug: 68Ga-Pentixafor

INTERVENTIONS:
Drug: 68Ga-Pentixather — After intravenous injection of 68Ga-pentixather, PET/CT scan will be performed.
  Other Names: 68Ga-Pentixather injection
Drug: 68Ga-Pentixafor — After intravenous injection of 68Ga-pentixafor, PET/CT scan will be performed.
  Other Names: 68Ga-Pentixafor injection

SUMMARY:
Chemokine receptor-4 (CXCR4) is overexpressed in multiple myeloma (MM) cells. 68Ga-pentixafor is a radio-labled tracer for CXCR4 . 68Ga-pentixafor PET/CT has shown good diagnostic performance in MM. But an exchange of Ga3+ by Lu3+ or Y3+ will lead to a significant loss of CXCR4 affinity. Investigators conduct this prospective study to evaluate the diagnostic performance of 68Ga-pentixather compared with 68Ga-pentixafor, in order to parallel 68Ga-pentixather and 177Lu/90Y-pentixather in theranostics of MM.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder which is characterized by clonal proliferation of plasma cell in bone marrow microenvironment. Chemokine receptor-4 (CXCR4) is overexpressed in MM cells, and has been identified as a potential therapy target. 68Ga-pentixafor is a radiolabeled ligand with high affinity for CXCR4. 68Ga-pentixafor PET/CT has been reported with better diagnostic performance than 18F-FDG PET/CT. However, considering both diagnostic and therapeutic applications, an exchange of Ga3+ by other M3+ ions (Lu or Y) will lead to a significant loss of CXCR4 affinity. Thus, pentixather was developed as the precursor of 177Lu-pentixather or 90Y-pentixather, which can be used in CXCR4-targeted peptide receptor radionuclide therapy (PRRT). Investigators conduct this prospective study to evaluate the diagnostic performance of 68Ga-pentixather compared with 68Ga-pentixafor, in order to parallel 68Ga-pentixather and 177Lu/90Y-pentixather in theranostics of MM.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or confirmed untreated multiple myeloma (MM), relapsed MM, MM in remission
2. Signed written consent

Exclusion Criteria:

1. pregnancy
2. breastfeeding
3. known allergy against pentixather or pentixafor
4. any medical condition that in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Metabolic parameter | through study completion, an average of 2 years
  Comparison of metabolic parameter (SUVmax) between 68Ga-pentixather PET/CT and 68Ga-pentixafor PET/CT.
PET-positive diffuse bone marrow involvement | through study completion, an average of 2 years
  Comparison of the number of diffuse bone marrow involvement between 68Ga-pentixather PET/CT and 68Ga-pentixafor PET/CT.
PET-positive focal bone marrow lesions | through study completion, an average of 2 years
  Comparison of the number of focal bone marrow lesions between 68Ga-pentixather PET/CT and 68Ga-pentixafor PET/CT.
PET-positive extramedullary lesions | through study completion, an average of 2 years
  Comparison of the number of extramedullary lesions between 68Ga-pentixather PET/CT and 68Ga-pentixafor PET/CT.

SECONDARY OUTCOMES:
Adverse effects | through study completion, an average of 2 years
  Types of adverse events.
Tumor burden assessment | through study completion, an average of 2 years
  The correlation between metabolic parameter (SUVmax) in 68Ga-pentixather PET/CT and clinical staging
Follow-up assessment | through study completion, an average of 2 years
  The correlation between metabolic parameter (SUVmax) in 68Ga-pentixather PET/CT and follow-up parameter (PFS).
CXCR4 expression in biopsies and metabolic parameters in PET | through study completion, an average of 2 years
  The correlation between CXCR4 expression in biopsies and metabolic parameter (SUVmax) in PET.

CONTACTS AND LOCATIONS:
Overall Officials: Qiao Yang, MD., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China